CLINICAL TRIAL: NCT02663024
Title: Phase 2, Randomized, Double-blind, Active-controlled, Dose-ranging Study to Evaluate the Pharmacokinetics, Pharmacodynamics and Safety of Idursulfase-beta (GC1111) in Hunter Syndrome (Mucopolysaccharidosis II) Patients
Brief Title: Study of Idursulfase-beta (GC1111) in Hunter Syndrome
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Green Cross Corporation (Industry)
Responsible Party: Sponsor
Organization: GC Biopharma Corp (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GC1111B_P2
Record Dates: First submitted 2016-01-17; First posted 2016-01-26 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Mucopolysaccharidosis II
MeSH Terms: conditions — Mucopolysaccharidosis II | interventions — idursulfase beta, mouse; idursulfase

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- Arm 1 (Experimental): 0.5 mg/kg, iv, weekly infusion of idursulfase beta for 24 weeks
  Interventions: Biological: idursulfase beta
- Arm 2 (Experimental): 1.0 mg/kg, iv, weekly infusion of idursulfase beta for 24 weeks
  Interventions: Biological: idursulfase beta
- Arm 3 (Experimental): 1.5 mg/kg, iv, weekly infusion of idursulfase beta for 24 weeks
  Interventions: Biological: idursulfase beta
- Arm 4 (Active Comparator): 0.5mg/kg, iv, weekly infusion of idursulfase for 24 weeks
  Interventions: Biological: idursulfase

INTERVENTIONS:
Biological: idursulfase beta — IV, weekly infusion for 24 weeks
  Other Names: GC1111
  Arms: Arm 1; Arm 2; Arm 3
Biological: idursulfase — 0.5 mg/kg, iv, weekly infusion for 24 weeks
  Other Names: Elaprase
  Arms: Arm 4

SUMMARY:
This study evaluates the efficacy and safety of three doses of GC1111 in patients with Hunter Syndrome. Participants will be randomized to one of three doses of GC1111 or comparator.

DETAILED DESCRIPTION:
This is a randomized, double-blind, active-controlled, dose-ranging study, where patient will receive one of the three doses of GC1111 (0.5 mg/kg, 1.0 mg/kg, and 1.5 mg/kg) or ELAPRASE 0.5 mg/kg. Approximately 20 patients will be administrated each study drug once every week as an iv infusion for 24 weeks. Efficacy of GC1111 will be evaluated in Six-Minute Walk Test (6MWT), urine Glycosaminoglycans(uGAG), liver and spleen volume, percent predicted Forced Vital Capacity(FVC), and cardiac size and function. Also immunogenicity, Pharmacokinetics(PK) and safety will be evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Male patients between 5 and 35 years of age
* Informed consent form signed
* Patients diagnosed with hunter syndrome
* Previously untreated with an enzyme replacement therapy

Exclusion Criteria:

* History of tracheostomy, bone marrow transplant, or cord blood transplant
* Treatment with another investigational product within 30 days prior to the start of study drug
* Known hypersensitivity of any of the ingredients of study drug
* Patient with severe hunter syndrome who cannot perform 6MWT
* Female patients

Ages: 5 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 20 (Estimated)
Dates: Start 2016-12; Primary Completion 2019-12 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in urinary GAG(Glycosaminoglycans) at Week 25 | Baseline to Week 25

SECONDARY OUTCOMES:
Change from baseline in urinary GAG at Week 25 | Baseline to Week 25
Change from baseline in Six Minute Walk Test at Week 25 | Baseline to Week 25
Percent change from baseline in Six Minute Walk Test at Week 25 | Baseline to Week 25
Change from baseline in Liver volume at Week 25 | Baseline to Week 25
  Liver volume measured by MRI
Percent change from baseline in Liver volume at Week 25 | Baseline to Week 25
  Liver volume measured by MRI
Change from baseline in Spleen volume at Week 25 | Baseline to Week 25
  Spleen volume measured by MRI
Percent change from baseline in Spleen volume at Week 25 | Baseline to Week 25
  Spleen volume measured by MRI
Incidence of Adverse Events and Serious Adverse Events | Baseline to Week 25
Safety changes from baseline in clinical laboratory tests, physical examination and vital signs | Baseline to Week 25
Immunogenicity | Baseline to Week 25
  anti-drug-antibody
Pharmacokinetic profile - Area under the serum concentration time curve (AUClast) | 1 and 17 week
Pharmacokinetic profile - Maximum observed peak plasma concentration (Cmax) | 1 and 17 week
Pharmacokinetic profile - Time at which Cmax is observed (Tmax) | 1 and 17 week

IPD SHARING:
Plan to Share IPD: No